CLINICAL TRIAL: NCT06414733
Title: Phase Ib Active Immunotherapy Trial (Expansion) With a Combination of Two Chimeric (Trastuzumab-like and Pertuzumab-like) HER-2 B Cell Peptide Vaccine Emulsified in ISA 720 Adjuvant in Patients With Advanced Solid Tumors
Brief Title: HER-2 B Cell Peptide Vaccine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pravin T.P Kaumaya (Other)
Responsible Party: Sponsor-Investigator, Pravin T.P Kaumaya, Director Brown Center for Immuno-Oncology and Vaccine Immunotherapy, Indiana University
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-09138
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Breast Cancer; Metastatic Gastrointestinal Carcinoma; HER2-positive Breast Cancer; HER2-positive Gastric Cancer; EGFR Overexpression
Keywords: Phase I; Breast Cancer; GI Cancer
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms | interventions — mannide monooleate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HER-2 vaccine Breast (Experimental)
  Interventions: Biological: Combination of MVF-HER-2 (597-626) and MVF-HER-2 (266-296) emulsified with ISA 720
- HER-2 vaccine GI (Experimental)
  Interventions: Biological: Combination of MVF-HER-2 (597-626) and MVF-HER-2 (266-296) emulsified with ISA 720

INTERVENTIONS:
Biological: Combination of MVF-HER-2 (597-626) and MVF-HER-2 (266-296) emulsified with ISA 720 — Three intramuscular (IM) injections (separated by 21 days) of a mixture of two peptides {MVF-HER-2(597-626) and MVF-HER-2 (266-296)} vaccine emulsified in ISA 720 vehicle. The combined vaccine preparation consists of 1.5mg of each of the HER-2 vaccine emulsified with a Montanide ISA 720, and will be administered in a final volume of 1.0 ml. Patients may also receive 6 months booster shots.

SUMMARY:
This phase I trial studies the side effects and best dose of vaccine therapy in treating patients with metastatic solid tumors. Vaccines made from antibodies and peptides combined with tumor cells may help the body build an effective immune response to kill tumor cells.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Extension and Expansion Cohorts

1. For the extension cohort to be conducted at the IUSCCC (N=12), patients with histologically documented metastatic or unresectable breast or gastrointestinal cancer will be enrolled.
2. For the expansion cohort (N=30), patients with either histologically documented metastatic or unresectable breast cancer (N=15), or histologically documented metastatic or unresectable gastrointestinal cancer (N=15) be enrolled. All patients enrolled to this cohort are required to have measurable disease. Note: Measurable disease is defined as ≥ 1 lesions that can be accurately measured in ≥ 1 dimensions as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan.

   Inclusion Criteria for all Cohorts:
3. Patients must have received or refused first line standard systemic therapy for their metastases (if applicable) and patients with histologically confirmed pancreatic and esophageal cancers must have received no more than two prior cytotoxic chemotherapy regimens in the last two years after standard therapy. Patients with histologically confirmed breast, and gastrointestinal cancers must have received no more than three prior cytotoxic chemotherapy regimens in the last two years after standard therapy.
4. Progressive disease after at least one line of standard therapy.
5. Patients with pancreatic and esophageal cancers must have received no more than two prior cytotoxic chemotherapy regimens in the last two years. Patients with breast and gastrointestinal cancers must have received no more than three prior cytotoxic chemotherapy regimens in the last two years.
6. Patients are required to have HER-2 (IHC 1+, 2+ and 3+) or EGFR over-expression (FISH and IHC) to be enrolled on this study.

   1. If the patient has had HER-2 expression measured prior to enrollment, the report alone will be accepted on the expansion phase of the study.
   2. If the patient has had EGFR expression measured prior to enrollment, the report alone will be accepted on the dose escalation phase of the study.
   3. If the patient has not had HER-2 or EGFR expression measured prior to enrollment on this study, it would be obligatory for the patient to have the tests performed to justify their status. HER-2 status can be performed by a variety of tests. Either IHC or FISH assay are acceptable if breast tumor tissues (previously frozen) are available. The test can be done at IUSCCC or elsewhere if the patient is from out of town.
7. Patients with prior history of treated brain metastases who are off steroids and have stable metastatic brain disease for at least 3 months are eligible.
8. Patients must be ambulatory with an ECOG performance status 0, 1, or 2 (appendix II).
9. Patients must have adequate organ function as defined by:

   1. ANC ≥ 1,000/mm³, platelet count > 700,000/mm³.
   2. Serum bilirubin < 1.5 mg%, regardless of whether patients have liver involvement secondary to tumor. ALT must be < 2 times upper limit of normal.
   3. Creatinine <1.5 mg/dl or calculated creatinine clearance > 60 ml/min
10. Patients must be at least 3 weeks past any prior surgery, cytotoxic, chemotherapy, other immunotherapy, hormonal therapy, or radiation therapy. Patients having been treated with monoclonal antibodies may enter the trial after a specified period of time (2 times the mean half life of the agent). Patients must have recovered from any toxicity of prior therapy prior to enrolling on study except for neuropathy where patients need to recover to less than grade 2.

    1. Patients with hormone receptor positive breast cancer who are on stable endocrine therapy are eligible if their tumor has some expression of HER-2 based on IHC of 1+ or 2+.
11. Patients must be at least 18 years of age.
12. Women of child-bearing potential must not be pregnant and must have a negative pregnancy test (Women of childbearing potential definition: (ECOG definition)).
13. Men and women must agree to practice effective contraception while on this study.
14. Patients must obtain a base line Echocardiogram or MUGA and require the left ventricular ejection fraction to be within normal limits (or 50% or higher).
15. Ability to understand and the willingness to sign a written informed consent document.

The patient must be aware that his/her disease is neoplastic in nature and willingly consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.

Exclusion Criteria:

1. Patients with tumors that are negative for HER-2 expression based on IHC of 0 AND Fluorescence in-situ hybridization showing lack of HER-2 amplification based on most recent ASCO/CAP guidelines; or are under-expressing EGFR based on FISH and IHC.
2. Patients on targeted therapies, such as Cycline Dependent Kinase (CDK) 4/6 or mammalian target of rapamycin (mTOR) inhibitors in combination with endocrine therapy
3. Patients who are {MVF-HER-2(266-296) and MVF-HER-2 (597-626)} immediate hypersensitivity skin test positive.
4. Patients who have evidence of active infection that requires antibiotic therapy. Patients must have been off antibiotic treatment for at least 3 weeks prior to initiating treatment and must be confirmed to be clear of the infection.
5. Patients with known active HIV, hepatitis A, hepatitis B, or hepatitis C infection.
6. Patients with serious uncontrolled cardiopulmonary disorders, including congestive heart failure, symptomatic coronary artery disease, serious cardiac arrhythmia, and symptomatic chronic obstructive pulmonary disease or patients with other serious uncontrolled medical diseases. At the discretion of the treating physician, patients who show disease control for at least 6 months may be enrolled.
7. Patients who require or likely to require corticosteroids or other immunosuppressives for intercurrent disease are NOT eligible.
8. Splenectomized patients.
9. Patients with active autoimmune diseases including rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis dermato-myositis, or a vasculitic syndrome.

   Note: At the discretion of the treating physician, patients who show disease control for at least 6 months may be enrolled.
10. Patients who have developed anaphylactic responses to other vaccines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety and toxicity at regular intervals by NCI common toxicity criteria 4.0 | through study completion (i.e. up to 1 year post initial vaccine)
Humoral Immune Response | through completion of 3 vaccine series (i.e. up to day 92 post final vaccine injection)
  Humoral immune response will be measured by ELISA quantification of IgM and IgG antibodies to HER2 (597-626) and HER2 (266-296)
Overall Response Rate | through completion of 3 vaccine series (i.e. up to day 71)

SECONDARY OUTCOMES:
immunogenicity | through study completion (i.e. up to 1 year post initial vaccine)
  ELISA will be analyzed for immunogenicity at baseline, with every vaccine, 21 days after the final vaccine, 6 months from initial vaccination, and at 1 year from initial vaccination to describe time course of antibody production
T cell functionality | through study completion (i.e. up to 1 year post initial vaccine)
  T cell functionality will be determined using proteomic profiling and immunophenotyping

CONTACTS AND LOCATIONS:
Overall Officials: Pravin Kaumaya, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Comprehensive Cancer Center, Indianpolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No